CLINICAL TRIAL: NCT03734315
Title: Routine Application of Ostenil® in Patients with Gonarthrosis
Status: Completed | Type: Observational
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Other Study IDs: OSTK-PMCF-DE-2018-01
Record Dates: First submitted 2018-10-30; First posted 2018-11-07 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ostenil®: 3-5 injections of sodium hyaluronate 1 % (20 milligrams (mg) / 2.0 millilitres (ml)) in weekly interval.
  Interventions: Device: Ostenil®

INTERVENTIONS:
Device: Ostenil® — Ostenil® is a CE-certified viscoelastic solution for injection into the joint cavity, containing 1.0 % sodium hyaluronate from fermentation.

SUMMARY:
PMCF study to observe the routine application of Ostenil® in the treatment of pain and restricted mobility in degenerative and traumatic changes of the knee joint.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age and in good general health condition
* Signed informed consent
* Existing Ostenil® recommendation for the treatment of gonarthrosis

Exclusion Criteria:

* Known hypersensitivity to one of the Ostenil® components
* Presence of articular effusion in study-relevant knee joint
* Known pregnancy or lactating females
* Subjects not capable of contracting and of understanding the nature, risks, significance and implications of the clinical investigation and unable to form a rational intention in the light of these facts
* Subjects unable to understand informed consent or having a high probability of non compliance to the study procedures and / or non completion of the study according to investigator's judgement (e.g. illiteracy, insufficient knowledge of local language)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 with Gonarthrosis and a Recommendation for Treatment with Ostenil®.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Change of Pain Intensity compared to Baseline (VAS-slider) | Day 7, Day 14, Day 21, Day 28, Day 84, Day 168, Day 252
  Evaluation of Pain Intensity by the Patient on a 10 cm VAS-slider. 10 cm equals the worst pain.
Change of Range of Motion compared to Baseline (Goniometer measurement) | Day 7, Day 14, Day 21, Day 28, Day 84, Day 168
  Assessment of the Range of Extension and Flexion of the Knee Joint using a Goniometer.
Change of Subjective Therapy Evaluation (KOOS Questionnaire) compared to Baseline | Day 84, Day 168
  Knee injury and Osteoarthritis Outcome Score (KOOS) to assess Stiffness, Pain, Function (daily living) and Quality of Life on a 5-point Likert scale.
Change of Subjective Symptom Evaluation (Overall Impression on a scale from 1 to 5) | Day 7, Day 14, Day 21, Day 28, Day 84, Day 168, Day 252
  The Change of Overall Subjective Symptom Evaluation on a scale from 1 (much improved) to 5 (much worse).
Incidence of Treatment-Emergent Adverse Events | Up to Day 252

CONTACTS AND LOCATIONS:
Overall Officials: Michael Krüger-Franke, Dr. med., Principal Investigator — MVZ am Nordbad
Locations (6):
- Germany (6):
  - Orthopädisches Versorgungszentrum München-Ost, Munich, Bavaria
  - Orthopädie am Altheimer Eck, München, Bavaria
  - Orthopädie München, München, Bavaria
  - Orthopädische Praxis am Isartor, München, Bavaria
  - MVZ am Nordbad, München, Bavaria
  - Orthopädische Praxis, München, Bavaria

IPD SHARING:
Plan to Share IPD: No